CLINICAL TRIAL: NCT01111149
Title: Varenicline and Smoking Cessation in Schizophrenia
Acronym: VSCS
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Double | Purpose: Treatment
Other Study IDs: 0904M64601; R01DA024674 (NIH)
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Results first posted 2014-07-03 (Estimated); Last update posted 2014-07-17 (Estimated); Status verified 2014-07

CONDITIONS: Schizophrenia; Smoking Cessation
Keywords: Schizophrenia; Smoking cessation; Varenicline; Bupropion
MeSH Terms: conditions — Schizophrenia; Smoking Cessation | interventions — Sugars; Varenicline; Bupropion

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Sugar Pill (Placebo Comparator): Sugar pill will be given to patients as a comparison group to the active varenicline group. In the fist week, one placebo pill will be given per patient, followed by 2 pills per day for the remaining 12 weeks of the study.
  Interventions: Other: Sugar Pill
- Varenicline (Experimental): Varenicline has not previously been examined for its efficacy and safety in subjects with schizophrenia. Subjects in the varenicline group will receive one 1mg pill/day for week 0, followed by two 1mg pills/day for the rest of the study. This is an experimental group to be compared against both placebo and bupropion HCl.
  Interventions: Drug: Varenicline
- Bupropion HCl (Active Comparator): Bupropion HCl is an established smoking cessation agent and will be used to compare its efficacy and safety against varenicline. Subjects in the Bupropion HCl group will receive one 150mg pill/day for week 0, followed by two 150mg pills/day for the rest of the study.
  Interventions: Drug: Bupropion HCl

INTERVENTIONS:
Other: Sugar Pill — Sugar pill created and masked by the pharmacy to be used as a control.
  Arms: Sugar Pill
Drug: Varenicline — Subjects in the varenicline group will receive one 1mg pill/day for week 0, followed by two 1mg pills/day for the rest of the study.
  Other Names: Chantix
  Arms: Varenicline
Drug: Bupropion HCl — in the Bupropion HCl group will receive one 150mg pill/day for week 0, followed by two 150mg pills/day for the rest of the study
  Other Names: Wellbutrin; Zyban
  Arms: Bupropion HCl

SUMMARY:
There is a strong association between smoking and schizophrenia with prevalence rates ranging from 74% to 90%, versus a national average of 30% in nonschizophrenic individuals. A number of hypotheses have been proposed to explain the relationship between high smoking rates and schizophrenia, mostly relating to self-medication primarily for the negative symptoms of schizophrenia. Smoking cessation rates among schizophrenic patients are considerably lower than for other psychiatric disorders. The negative health effects of smoking increase the morbidity and mortality in schizophrenic patients. Currently, the efficacy of bupropion HCl in the treatment of smoking by schizophrenic subjects is inconclusive, and there have not been any published studies of the efficacy of varenicline in schizophrenic subjects. As varenicline appears to be a promising treatment in non-psychiatric patients, it would be useful to expand these studies to examine its effects in schizophrenic patients. Identifying effective and safe means of smoking cessation for this vulnerable population has the potential to reduce morbidity and mortality among individuals with schizophrenia.

DETAILED DESCRIPTION:
There is a strong association between smoking and schizophrenia with prevalence rates ranging from 74% to 90%, versus a national average of 30% in nonschizophrenic individuals. A number of hypotheses have been proposed to explain the relationship between high smoking rates and schizophrenia, mostly relating to self-medication primarily for the negative symptoms of schizophrenia. Smoking cessation rates among schizophrenic patients are considerably lower than for other psychiatric disorders. The negative health effects of smoking increase the morbidity and mortality in schizophrenic patients. The smoking cessation agent bupropion HCl has been tested in schizophrenics, but the results on its efficacy are inconclusive. Recent works by different laboratories have shown the safety and efficacy of varenicline, a partial alpha4beta2 and full alpha7 nicotinic acetylcholine receptor agonist, as a smoking cessation agent. However, to date, no published studies have tested the safety and efficacy of varenicline in treatment of nicotine dependence in schizophrenic patients. As varenicline appears to be a promising treatment in non-psychiatric patients, it would be beneficial to examine its effects in schizophrenic patients. The central hypothesis of this application is that treatment with varenicline will safely increase smoking abstinence rates in schizophrenic patients when compared to those receiving placebo. This central hypothesis will be tested and the objectives of this application accomplished by pursuing two Specific Aims: 1) Treatment with varenicline or bupropion HCl for a period of three months will increase smoking abstinence rates in schizophrenic patents when compared to placebo; and 2) Treatment with varenicline or bupropion HCl for a period of three months will not increase psychosis in schizophrenic patients when compared to placebo. For our General Investigational Plan, we will employ a double-blind randomized placebo controlled study to assess varenicline's safety and efficacy. It is our expectation that we will demonstrate that varenicline is safe and effective in decreasing smoking rates in schizophrenic patients without exacerbating psychotic symptoms. Such outcomes will be significant, because they will offer a new treatment for smoking cessation in this vulnerable population.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects, 18-75 years old
* Diagnosis of schizophrenia or schizoaffective disorder based on Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria
* Smoking at least 10 cigarettes per day
* Weight of at least 100 lbs (45.4 kg)
* Motivation to quit smoking
* Stabilized psychotic symptoms
* Provision of informed consent for testing and treatment

Exclusion Criteria:

* Serious cardiac, renal, hypertensive, pulmonary, endocrine, or neurologic disorder
* Seizure disorder, recent withdrawal from alcohol or anxiolytics
* History of bulimia nervosa, anorexia nervosa, or dementia
* History of depression, panic, or bipolar disorders
* Pregnancy or lactation
* Prior use of varenicline or bupropion HCl within three months prior to initiation of the study
* Current use of other smoking cessation treatments
* Regular use of non-cigarette tobacco products (> than once/week)
* Past substance abuse (alcohol or non-nicotine containing drugs) in the preceding 6 months
* Patients with suicidal ideations or plans
* Florid psychosis or increasing psychosis following varenicline or bupropion HCl treatment
* History of, or current, alcohol dependence/abuse
* Current use of monoamine oxidase inhibitors (MAOI)

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2009-12; Primary Completion 2012-08 (Actual); Study Completion 2012-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: S. Hossein Fatemi, M.D., Ph.D., Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, University of Minnesota Medical Center, Minneapolis, Minnesota, United States

REFERENCES:
- [Background] Yousefi MK, Folsom TD, Fatemi SH. A Review of Varenicline's Efficacy and Tolerability in Smoking Cessation Studies in Subjects with Schizophrenia. J Addict Res Ther. 2011 Dec 20;S4(1):3045. doi: 10.4172/2155-6105.S4-001. PMID 22514788
- [Background] Fatemi SH. Varenicline efficacy and tolerability in a subject with schizophrenia. Schizophr Res. 2008 Aug;103(1-3):328-9. doi: 10.1016/j.schres.2008.05.002. Epub 2008 Jun 24. No abstract available. PMID 18572388
- [Result] Fatemi SH, Yousefi MK, Kneeland RE, Liesch SB, Folsom TD, Thuras PD. Antismoking and potential antipsychotic effects of varenicline in subjects with schizophrenia or schizoaffective disorder: a double-blind placebo and bupropion-controlled study. Schizophr Res. 2013 May;146(1-3):376-8. doi: 10.1016/j.schres.2013.02.015. Epub 2013 Mar 16. No abstract available. PMID 23507358
- [Derived] Livingstone-Banks J, Fanshawe TR, Thomas KH, Theodoulou A, Hajizadeh A, Hartman L, Lindson N. Nicotine receptor partial agonists for smoking cessation. Cochrane Database Syst Rev. 2023 May 5;5(5):CD006103. doi: 10.1002/14651858.CD006103.pub8. PMID 37142273

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 12/15/2009 through 4/03/2012. Fliers advertising the study were placed in medical clinics. Additionally, advertisements were placed in local newspapers City Pages and The Minneapolis Star Tribune.
Pre-assignment Details: Enrolled participants were excluded from the trial before assignment to groups if they no longer showed interest in the study or failed drug screens.
Period: Overall Study
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Started | 9 | 6 | 9
Completed | 7 | 5 | 5
Not Completed | 2 | 1 | 4
Not completed — Protocol Violation | 1 | 1 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl | Total
Number analyzed (Participants) | 9 | 6 | 9 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.4 (9.8) | 40.4 (15.9) | 43 (8.44) | 41.46 (11.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 1 | 2 | 5
  Male | 7 | 5 | 7 | 19
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 3 | 2 | 6
  White | 8 | 3 | 6 | 17
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 9 | 6 | 9 | 24
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 9 | 6 | 9 | 24

OUTCOME MEASURES:

1. Primary Outcome: Smoking Abstinence - Serum/Urine Measurements
Description: Measured by blood/urine tests for nicotine and its break-down product cotinine.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
ng/mL
  Serum Cotinine (Week 12) | 198.67 (129.84) | 207 (130.73) | 213.8 (137.6)
  Serum Nicotine (Week 12) | 22.57 (24.23) | 6 (9.59) | 15.4 (11.61)
  Urine Cotinine (Week 12) | 772 (381.19) | 699.6 (527.45) | 614.75 (469.54)
  Urine Nicotine (Week 12) | 820 (301.46) | 613.25 (243.29) | 412.75 (487.9)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for Serum Cotinine at Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for Serum Nicotine at Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for Urine Cotinine at Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for Urine Nicotine at Week 12; Test type: Superiority or Other; p > 0.05, ANOVA

2. Secondary Outcome: Reduction in Smoking
Description: Successful outcome will be defined as a 50% or greater reduction in self-reported cigarettes per day and a 30% greater reduction in carbon monoxide and cotinine levels. Measured at week 12
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
participants
  50% Reduction in Number of Cigarettes Smoked | 2 | 2 | 1
  30% Reduction in Carbon Monoxide (Week 12) | 2 | 2 | 1
  30% Reduction in Serum Cotinine (Week 12) | 2 | 4 | 1
  30% Reduction in Urine Cotinine (Week 12) | 2 | 4 | 1
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for 50% Reduction in Number of Cigarettes Smoked (Week 12); Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for 30% Reduction in Carbon Monoxide (Week 12); Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for 30% Reduction in Serum Cotinine (Week 12); Test type: Superiority or Other; p > 0.05, Chi-squared
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for 30% Reduction in Urine Cotinine (Week 12); Test type: Superiority or Other; p > 0.05, Chi-squared

3. Secondary Outcome: Negative Symptoms of Schizophrenia - SANS
Description: Scale for the Assessment of Negative Symptoms (SANS) a well-established test, used to assess the presence of psychosis or negative symptoms of schizophrenia. It consists of 25 questions rated on a scale of 0 (none) to 5 (severe). With a total score range of 0 to 125 points. There are 6 subscales: Affective Flattening or Blunting - (minimum, 0; maximum 35); Inappropriate Affect (minimum, 0; maximum 5); Alogia (minimum 0; maximum 25); Avolition-Apathy (minimum 0; maximum 20); Anhedonia-Asociality (minimum 0; maximum 25); Attention (minimum 0; maximum 15). Each subscale (except for Inappropriate Affect) contains one additional question as a Global Rating - or overall measure for that particular subscale. The sum of these questions constitutes the Total Global Score (minimum 0, maximum 25). The global questions are included within the Total Composite score. In each case, the larger the score, the more severe the symptoms.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  SANS Total Composite (Week 12) | 5.86 (5.24) | 17.2 (9.83) | 6.20 (5.12)
  SANS Total Global (Week 12) | 1.71 (1.50) | 3.8 (2.49) | 1.6 (1.82)
  SANS Affective Flattening (Week 12) | 1.57 (3.36) | 7 (3.81) | 0.8 (1.10)
  SANS Alogia (Week 12) | 0.71 (1.89) | 0.6 (1.34) | 0 (0)
  SANS Avolition (Week 12) | 2 (2.77) | 3 (3.67) | 3.6 (3.78)
  SANS Anhedonia (Week 12) | 1.57 (1.99) | 5.8 (7.36) | 1.4 (3.13)
  SANS Attention (Week 12) | 0 (0) | 0.2 (0.45) | 0 (0)
  Inappropriate Affect (Week 12) | 0 (0) | 0.60 (0.88) | 0.40 (0.89)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Total Composite (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Total Global (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Affective Flattening (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Alogia (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Avolition (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Anhedonia (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 7: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SANS Attention (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 8: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis of Inappropriate Affect at Week 12; Test type: Superiority or Other; p > 0.05, ANOVA

4. Secondary Outcome: Impulsivity and Inattention
Description: Impulsivity and inattention will be measured using the continuous performance test. Individuals were tasked with 359 items divided six blocks (59 in block 1, 60 in blocks 2-6). Omissions result from the failure to respond to target letters. CPT% Omissions measures the percentage of responses that qualify as omissions made during the test. Higher scores indicate increased inattention. Commissions result from responses given to non-targets. CPT% Commissions measures the percentage of responses that qualify as commissions made during the test. Higher scores indicate increased inattention. Perseverations result from reaction time less than 100 ms. CPT% Perseveration % measures the percentage of responses that qualify as perseverations made during the test. The higher the score, the greater impulsivity.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: Percentage of responses
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
Percentage of responses
  CPT % Omissions (Week 12) | 5.62 (11.14) | 0.68 (1.04) | 2.42 (2.66)
  CPT % Commissions (Week 12) | 36.11 (22.64) | 25 (37.89) | 28.33 (21.82)
  Perseveration % (Week 12) | 0.57 (0.86) | 1.05 (1.84) | 0.12 (0.17)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for CPT % Omissions (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for CPT% commissions (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for perseveration % (week 12); Test type: Superiority or Other; p > 0.05, ANOVA

5. Secondary Outcome: Side Effects
Description: Side effects will be monitored by a physician and/or assistant and recorded (SEP). All patients withdrawn from the study because of emerging side effects will be followed until the side effects are resolved. Each item is scored based on a scale of 0=none; 1=mild; 2=moderate; and 3=severe. Below, the data are shown for participants experiencing symptoms on week 12 of the study.
Time Frame: Week 12
Measure: Number; unit: participants
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
participants
  Anxiety | 3 | 3 | 0
  Dizziness | 0 | 0 | 1
  Mania | 0 | 0 | 0
  Abnormal Dreams | 3 | 1 | 0
  Abdominal Pain | 0 | 1 | 1
  Headache | 3 | 3 | 0
  Insomnia | 1 | 0 | 1
  Nausea | 0 | 2 | 1
  Psychosis | 0 | 0 | 1
  Dry Mouth | 2 | 0 | 0
  Chest Pain | 0 | 0 | 0
  Irregular Heart Beat | 0 | 0 | 0
  Weakness/Fainting | 2 | 0 | 1
  Diarrhea | 1 | 1 | 0
  Vomiting | 0 | 0 | 0
  Constipation | 0 | 1 | 1
  Confusion | 0 | 1 | 1
  Irritability | 1 | 0 | 1
  Drooling | 0 | 1 | 1
  Cold Sweats | 0 | 0 | 0
  Blurred Vision | 0 | 1 | 1
  Leg Pain/Cramps | 2 | 1 | 0
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Anxiety at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Dizziness at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Mania at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for abnormal dreams at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 5: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Abdominal Pain at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 6: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Headache at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 7: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Insomnia at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 8: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Nausea at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 9: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Psychosis at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 10: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Dry Mouth at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 11: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Chest Pain at Week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 12: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Irregular Heart Beat at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 13: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Weakness/Fainting at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 14: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Diarrhea at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 15: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Vomiting at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 16: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Constipation at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 17: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Confusion at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 18: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Irritability at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 19: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for drooling at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 20: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Cold Sweats at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 21: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Blurred Vision at week 12; Test type: Superiority or Other; p > 0.05, Fisher Exact
Statistical Analysis 22: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Leg Pain/Cramps; Test type: Superiority or Other; p > 0.05, Fisher Exact

6. Secondary Outcome: Abstinence-related Symptoms - MNWS and FTND
Description: Minnesota Nicotine Withdrawal Scale (MNWS), a patient-reported measure of nicotine withdrawal symptoms and cravings. Eight items are listed, including craving for cigarettes, irritability, frustration, or anger, anxiety, etc scored on a five point scale from 0 (normal) to 5 (severe). Patients are asked for responses for the past 24 hours and past seven days (minimum 0, maximum 32; for each subscale). The higher the score, the greater the dependence. Additionally, one question (minimum score 1, maximum score 4 measures the individual's confidence in resisting strong urges to smoke. The higher the score on this question, the greater the individual's confidence in resisting smoking urges.
  The Fagerstrom Test for Nicotine Dependence measures nicotine dependence and consists of six questions with a total minimum score of 0 and a maximum score of 10. The higher the score, the greater the dependence on nicotine.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  FTND (Week 12) | 4.86 (1.77) | 5.2 (1.48) | 4.4 (3.36)
  MNWS 24 Hour Total (Week 12) | 7.29 (7.04) | 8.2 (7.36) | 6.60 (4.67)
  MNWS 7 day total (Week 12) | 9.14 (4.98) | 11 (4.64) | 5.80 (4.27)
  MNWS Resistance (Week 12) | 2.71 (1.11) | 3.4 (0.55) | 2.4 (1.14)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for FTND (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for MNWS 24 Hour Total (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for MNWS 7 day total (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for MNWS Resistance (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

7. Secondary Outcome: Depression
Description: Beck Depression Inventory (BDI), a self-report rating inventory measuring characteristic attitudes and symptoms of depression consisting of 21 items with each item rated on a four point scale (0=not present to 3=severe). The accepted ranges are as follows: 0 to 9 indicates no depression, 10 to 18 indicates mild to moderate depression, 19 to 29 indicates moderate to severe depression and 30 to 63 indicates severe depression.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale | 3.71 (3.55) | 8.6 (9.94) | 5.4 (6.99)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis of Beck Depression Inventory (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

8. Secondary Outcome: Abnormal Movements - BAS and SAS
Description: Barnes Akathisia Scale (BAS), a widely-used measurement of drug-induced akathisia. It consists of 4 questions with questions 1-3 scored on a scale of 0-3 with 0=normal and 3=severe (minimum score 0, maximum score 9; while item 4 is a global clinical assessment of akathisia rated on a scale of 0 (normal) to 5 (severe). The higher the score on each subsclae, the greater the severity of akathisia.
  Simpson-Angus Scale (SAS), a 10-item instrument used to evaluate patients experiencing neuroleptic-induced parkinsonism and other extrapyramidal side effects. Items are rated for severity on a 0-4 scale, with 0 being normal and 4 being severe. Minimum = 0; Maximum = 40. The higher the score, the greater the severity.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  SAS (Week 12) | 0.2 (0.24) | 0.76 (0.76) | 0.42 (0.8)
  BAS Items 1-3 (Week 12) | 0.57 (0.98) | 0.6 (0.89) | 0.4 (0.89)
  BAS Item 4 (Week 12) | 0.29 (0.49) | 0.4 (0.55) | 0.2 (0.45)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SAS (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for BAS items 1-3 (week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for BAS item 4 (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

9. Secondary Outcome: Vital Signs
Description: blood pressure will be measured.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: mm Hg
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
mm Hg
  Systolic Blood Pressure (Week 12) | 116.29 (15.53) | 122 (7.34) | 128.4 (32.42)
  Diastolic Blood Pressure (Week 12) | 76.71 (9.94) | 78.4 (8.14) | 74.8 (10.71)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for systolic blood pressure (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for diastolic blood pressure (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

10. Secondary Outcome: Vital Signs - Weight
Description: Weight will be measured for each participant. Values listed below are for week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: lbs
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
lbs | 218.39 (69.64) | 213.47 (35.2) | 254.78 (65.50)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Vital Signs - Weight (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

11. Primary Outcome: Smoking Abstinence - Number of Cigarettes Smoked
Description: Number of cigarettes smoked at week 12 of the study by self-report.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: number of cigarettes smoked
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
number of cigarettes smoked | 19.71 (22.77) | 9.4 (5.47) | 17.1 (17.28)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Smoking Abstinence - Number of Cigarettes Smoked (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

12. Primary Outcome: Smoking Abstinence - Exhaled Carbon Monoxide
Description: Exhaled carbon monoxide as a biochemical verification of smoking abstinence. Values below are for week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: parts per million
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
parts per million | 21.14 (18.51) | 17 (13.53) | 22.6 (19.14)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Smoking Abstinence - Exhaled Carbon Monoxide (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

13. Secondary Outcome: Vital Signs - Pulse
Description: Pulse will be measured. The values below were measured at week 12 of the study.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: heart beats per minute
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
heart beats per minute | 82.57 (15.76) | 87 (13.43) | 89.2 (18.47)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Vital Signs - Pulse (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

14. Secondary Outcome: Suicidality
Description: The Columbia-Suicide Severity Rating Scale (C-SSRS), is a survey intended to quantify the severity of suicidal ideation and behavior. The questionaire for suicidal ideation consists of 5 questions with yes (1) /no (0) answers. If answers to questions 1 and 2 are no, questions 3-5 are skipped. Minimum of 0; Maximum of 5. The questionaire for suicidal behavior consists of seven questions rated 0 for no and 1 for yes. The minimum score is 0 and the maximum score is 7. In each case, the higher the score, the greater the severity.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  Lifetime Suicidal Ideation (week 12) | 1.71 (1.7) | 0.8 (0.84) | 0.4 (0.55)
  Lifetime Suicide Attempts (week 12) | 1.29 (1.7) | 1.2 (1.3) | 0.4 (0.55)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Lifetime Suicidal Ideation (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Lifetime Suicide Attempts (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

15. Secondary Outcome: Positive Symptoms of Schizophrenia (SAPS)
Description: Scale for the Assessment of Positive Symptoms (SAPS), a well-established test, used to assess the presence of psychotic symptoms of schizophrenia. There are 34 items rated on a scale of 0-5 with 0=none and 5=severe for a minimum score of 0 and a maximum score of 170. There are 4 subscales: Hallucinations (minimum score 0; maximum score 35); Delusions (minimum score 0; maximum score 65); Bizarre Behavior (minimum score 0; maximum score 25); Positive Formal Thought Disorder (minimum score 0; maximum score 45). Each subscale contains one additional question as a Global Rating - or overall measure for that particular subscale. The sum of these questions constitutes the Total Global Score (minimum 0, maximum 20). The values for the Global items are included in the Total Composite score. In each case, the higher the score, the greater the severity of symptoms.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  SAPS Total Composite Score - Week 12 | 3.43 (4.86) | 7 (7.48) | 10.6 (7.7)
  SAPS Total Global - Week 12 | 1.29 (1.89) | 1.2 (1.3) | 1.8 (1.3)
  SAPS Hallucinations - Week 12 | 2 (3.83) | 2.2 (2.59) | 3 (4.12)
  SAPS Delusions - Week 12 | 1.43 (1.9) | 4.2 (7.36) | 3.8 (3.56)
  SAPS Bizarre Behavior - Week 12 | 0 (0) | 0 (0) | 0.4 (0.55)
  SAPS Thought Disorder - Week 12 | 0 (0) | 0.6 (1.34) | 3.4 (5.64)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SAPS Total Composite Score - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline; Statistical analysis for SAPS Total Global - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SAPS Hallucinations - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Delusions - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for SAPS Bizarre Behavior - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for SAPS Thought Disorder - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA

16. Secondary Outcome: General Psychopathology
Description: Brief Psychiatric Rating Scale (BPRS), an 24-item scale measuring positive symptoms, general psychopathology, and affective symptoms commonly used for schizophrenia with each item rated on a scale of 1-7 with 1=not present and 7=severe. The minimum score is 24 and the maximum score is 168. We have used five subscales as recommended by Dingemans et al., 1995: Positive subscale (minimum score 6; maximum score 42); Negative subscale (minimum score 5; maximum score 35); Depressed subscale (minimum score 5; maximum score 35); Mania subscale (minimum score 6; maximum score 42); and Disorientation subscale (minimum score 2; maximum score 14) . For both the total score and the subscale scores, the higher the score, the greater the symptom severity. We used the BPRS version 4.0. Dingemans PMAJ, Linszen DH, Lenoir ME, Smeets RMW, 1995. Component structure of the expanded Brief Psychiatric Rating Scale (BPRS-E). Psychopharmacology 122:263-267.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  BPRS Total - Week 12 | 30 (4.47) | 34.2 (3.96) | 31.6 (4.28)
  BPRS Positive Subscale - Week 12 | 8.14 (2.73) | 9 (2.74) | 8 (2.92)
  BPRS Negative Subscale - Week 12 | 6 (1.15) | 6.4 (1.67) | 7.4 (1.52)
  BPRS Mania Subscale - Week 12 | 6.43 (1.13) | 6.4 (0.55) | 8 (2.92)
  BPRS Disorientation Subscale - Week 12 | 2 (0) | 2 (0) | 2 (0)
  BPRS Depression Subscale - Week 12 | 7.43 (2.64) | 10.4 (2.88) | 6.2 (1.79)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for BPRS Total - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for BPRS Positive Subscale - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for BPRS Negative Subscale - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 4: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Mania Subscale - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 5: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Disorientation Subscale - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 6: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for BPRS Depression Subscale - Week 12; Test type: Superiority or Other; p > 0.05, ANOVA

17. Secondary Outcome: Hit Reaction Time - CPT
Description: The hit reaction time is the average speed of correct responses for the entire test given in milliseconds. The higher the score, the slower the speed. The standard error is a measure of response speed consistency. The higher the overall standard error, the greater inconsistency in the response speed. The values below were measured at week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
milliseconds
  Hit Reaction Time (week 12) | 42.44 (36.91) | 67.61 (34.47) | 63.81 (41.80)
  Hit Reaction Time Standard Error (Week 12) | 7.20 (4.83) | 6.96 (2) | 8.79 (3.02)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Hit Reaction Time - CPT (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

18. Secondary Outcome: Variability of Standard Error - CPT
Description: Variability of Standard Error (VSE) is a measure of response speed consistency. VSE measures "within respondent" variability. That is, the amount of variability the individual shows in 18 separate segments of the Continuous Performance Test in relation to his or her own overall standard error. Although VSE is a different measure than Overall Standard Error, typically the two measures produce comparable results. The higher the VSE, the greater the inconsistency in the response speed. The values shown below are the VSE for Week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
milliseconds | 11.05 (10.99) | 11.38 (6.84) | 11.8 (6.01)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Variability of Standard Error - CPT (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

19. Secondary Outcome: Detectibility (d') of Continuous Performance Test
Description: The value d' is a measure of the difference between the signal (non-X) and noise (X) distributions. As such, d' provides a means for assessing an individual's discriminative power since, in general, the greater the difference between the signal and noise distributions, the better the ability to distinguish and detect X and non-X stimuli. The lower the score, the better the detectability. Values shown below are for week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: unitless
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
unitless | 0.71 (0.54) | 1.32 (0.80) | 1.09 (0.68)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Detectibility (d') of Continuous Performance Test (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

20. Secondary Outcome: Response Style Indicator (Beta) for CPT
Description: Beta represents an individual's response tendency: Some individuals are cautious and choose not to respond very often. Conceptually, such individuals want to make sure they are correct when they give a response. Higher values of Beta reflect this response style. The emphasis is on avoiding commission errors. Other individuals respond more freely to make sure they respond to most or all targets, and they tend to be less concerned about mistakenly responding to a non-target. Lower values of Beta are produced by this response style. Values shown below were obtained at week 12.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: Beta
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
Beta | 0.95 (0.55) | 1.41 (1.48) | 2.92 (4.13)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for Response Style Indicator (Beta) for CPT (week 12); Test type: Superiority or Other; p > 0.05, ANOVA

21. Secondary Outcome: Abstinence Related Symptoms - WISDM
Description: The Wisconsin Inventory of Smoking Dependence Motives (WISDM) consists of 68 items regarding smoking. Each item is rated on a scale of 1 (not true of me at all) to 7 (extremely true of me) leading to a minimum score of 68 and a maximum score of 476. The higher the score, the greater the dependence. Four of the items are grouped into a Craving subscale (minimum 4, maximum 28), the greater the score, the greater the craving. Five of the items are grouped into a Cognition subscale (minimum 5, maximum 35), the higher the score, the greater reliance on cigarette smoking for cognitive enhancement. WISDM scoring based on the original article by Piper et al., 2004. A multiple motives approach to tobacco dependence: the Wisconsin inventory of smoking dependence motives (WISDM-68). Journal of Consulting and Clinical Psychology 72:139-154.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  WISDM Total (Week 12) | 229.14 (93.31) | 229.4 (52.03) | 270.6 (181.21)
  WISDM Cognition (Week 12) | 11.57 (8.87) | 15.4 (5.81) | 23.2 (16.16)
  WISDM Craving (Week 12) | 15.14 (5.73) | 14.2 (3.35) | 18 (11.11)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for WISDM Total (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for WISDM Cognition (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for WISDM Craving (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

22. Secondary Outcome: Urge to Smoke - MNWS
Description: The Minnesota Nicotine Withdrawal Scale (MNWS) includes two items where individuals are asked to 1) declare the percentage of time they had an urge to smoke (MNWS % Urge to Smoke); and 2) declare the percentage of time they had a strong urge to smoke (MNWS % Strong Urge). For each case, percentages range from 0% to 100% - the higher the percentage, the greater urge to smoke.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
percentage of time
  MNWS % Urge to Smoke (Week 12) | 36.43 (18.87) | 47 (22.8) | 47 (34.21)
  MNWS % Strong Urge (Week 12) | 26.43 (23.4) | 33 (18.57) | 32.4 (40.61)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for MNWS % Urge to Smoke (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for MNWS % Strong Urge (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

23. Secondary Outcome: Abnormal Movements - AIMS
Description: Abnormal Involuntary Movement Scale (AIMS), to assess abnormal involuntary movements associated with antipsychotic drugs. There are 10 questions, based on a five-point scale ranging from 0 (none) to 4 (severe). Items 11-14 are yes/no questions that have no impact on the score. The Total Score is the sum of questions 1-7 (minimum = 0; maximum = 28). The severity index consists of one question (item 8; rated 0=none to 4=severe) based on the rater's observation of abnormal movements The AIMS Global Score is the sum of three questions (each item rated 0=none to 4=severe) regarding abnormal movements overall (minimum score 0, maximum score 12). For the total score and subscores, the higher the score, the greater the severity of abnormal movements. Scoring is based on the chapter: Guy W (2000), Abnormal Involuntary Movement Scale (AIMS), in: Handbook of Psychiatric Measures (Rush AJ Jr, et al., eds). APA Publishing: Washington DC: pp. 166-167.
Time Frame: Week 12
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Number analyzed (Participants) | 7 | 5 | 5
units on a scale
  AIMS Total (Week 12) | 0.71 (1.25) | 1 (1.41) | 1.40 (2.19)
  AIMS Severity Index (Week 12) | 0 (0) | 0.2 (0.45) | 0.4 (0.89)
  AIMS Global Score (Week 12) | 0 (0) | 0.2 (0.45) | 0.6 (1.34)
Statistical Analysis 1: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for AIMS Total (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 2: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical analysis for AIMS Severity Index (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA
Statistical Analysis 3: Comparison: Sugar Pill vs Varenicline vs Bupropion HCl; Statistical Analysis for AIMS Global Score (Week 12); Test type: Superiority or Other; p > 0.05, ANOVA

ADVERSE EVENTS:
Arm/Group | Sugar Pill | Varenicline | Bupropion HCl
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/7 | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No